CLINICAL TRIAL: NCT04427150
Title: Examining Affective Prosody Recognition Among Children With Autism Spectrum Disorders and the Effectiveness of an Auditory Intervention Using a Mobile App
Brief Title: Affective Prosody Recognition and Auditory Intervention for Children With Autism Spectrum Disorders (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: The Hong Kong Polytechnic University (Other); Education University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ming Lui, Associate Professor, Hong Kong Baptist University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKBU 12604418
Record Dates: First submitted 2020-06-01; First posted 2020-06-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: 120 participants (60 children with autism spectrum disorder and 60 typically developed children) will form three groups: Group 1 will contain 30 children with autism spectrum disorder (randomly selected) whom will partake in psychoacoustic intervention training. Group 2 will contain 30 children with autism spectrum disorder (randomly selected) whom will partake in non-psychoacoustic intervention training. Group 3 will contain 60 typically developed children whom will not partake in any training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auditory Training Group (Experimental): 12 hours of psychoacoustic training over 8 weeks
  Interventions: Behavioral: Auditory Training
- Other Training Group (Active Comparator): 12 hours of non-psychoacoustic training over 8 weeks
  Interventions: Behavioral: Non-auditory training
- TD Group (No Intervention)

INTERVENTIONS:
Behavioral: Auditory Training — A series of psychoacoustic training exercises through Posit Science - BrainHQ (mobile app or web-browser version). Each training is approximately 2 minutes
  Arms: Auditory Training Group
Behavioral: Non-auditory training — A series of non-psychoacoustic training exercises through Posit Science - BrainHQ (mobile app or web-browser version). Each training is approximately 2 minutes
  Arms: Other Training Group

SUMMARY:
The proposed study aims to examine the abilities of children with ASD to recognize emotional tones of voice - also known as affective prosody - as compared to typically developing (TD) children. Past findings are mixed, and although some studies have found intact performance among individuals with ASD, it is possible that they rely on different underlying mechanisms in processing affective prosody compared to TD children. Our second objective is therefore to examine whether children with ASD have a stronger reliance on psychoacoustic abilities - including rapid auditory processing and pitch direction recognition - to identify emotional stimuli, as compared to TD children. Lastly, the investigators will study whether auditory training targeting psychoacoustic abilities would improve affective prosody recognition among children with ASD. Sixty children with ASD and 60 TD children between 10 to 12 years old will be recruited. Participants' psychoacoustic abilities and affective prosody recognition will be assessed in the pretest. The investigators hypothesize that psychoacoustic abilities are stronger predictors of affective prosody recognition among children with ASD than among TD children. The ASD children will then be randomly assigned to two groups: one group will receive auditory training; the other will be an active control group that receives non-auditory training. Both groups will receive 12 hours of training via a mobile app. The children will be assessed again in the posttest.

DETAILED DESCRIPTION:
Participants will sign an informed consent statement prior to arriving at the lab. Participants with ASD will be randomly assigned into either the auditory training group (Group 1) or the active control group (Group 2). Participants without ASD will be assigned to the typically developed group (Group 3). Groups 1 and 2 will complete all stages of the study, whereas Group 3 will only complete the pre-test stage.

Pre-test: Researchers will assess participants' affective prosody recognition ability and psychoacoustic ability. The tests will be conducted in a sound attenuated lab located at Hong Kong Baptist University. The tests include an affective prosody recognition test, a pitch discrimination recognition test, a rapid auditory processing test, and a theory of mind test.

Intervention Training: Participants will be required to partake in an intervention training program. The program will adopt training exercises provided by Posit Science - BrainHQ. The participants will be asked to complete a training session of 15-30 minutes each day for 8 weeks, arriving at a total of at least 8 hours of training. The progress of intervention training will be closely monitored by the research team.

Post-test: Participant will be asked to return to the lab for post-test assessment of the same tests, and complete an autism assessment (ADOS-2) and intelligence assessment (WISC-IV) conducted by a clinical psychologist, as well as a non-verbal Intelligence test (KBIT-2) conducted by a trained researcher.

Note: For ethical and fairness purposes, participants from Group 2 will be allowed to access the intervention training after Post-test.

To encourage completion of the intervention training program, participants who successfully complete 8 hours of training will be offered a monetary reward as a token of appreciation.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese as mother language
* IQ > 70
* Children with autism spectrum disorder

Exclusion Criteria:

* Children diagnosed with dyslexia
* Prior diagnosis of mental disorders

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Accuracy of Affective Prosody Recognition | Before & after 8-week intervention program
  Measures the change in the participants' ability in identifying emotional tone of words or sentences (sound stimuli). The participant will be tested before intervention and after intervention. For each test, participants will listen to word or sentences, which are pre-recorded by voice actors, then identify the emotional tone (happy, anger, fear, sad, or neutral) of the stimuli by pressing the corresponding keys on the keyboard. The accuracy of response will be used to assess the participants' ability.
Change in Ability in Discriminating Pitch Differences | Before & after 8-week intervention program
  Measures the change the participants' ability in discriminating the pitch between two tones using the Pitch Discrimination Recognition task. The participant will be tested before intervention and after intervention. For each test, participants will listen to two tones and will be required to identify which tone has the higher pitch. The pitch difference between the two tones will change using a "two-down one-up" mechanism with a step-wise adjustment, which means the pitch difference will decrease every two consecutive correct responses or increase for every incorrect response. For every reversal (change from decrease to increase or vice versa) of stimuli, the latest pitch difference will be recorded. The average pitch difference of the final 8 reversals will be used to assess the participants' pitch discrimination ability. Lesser difference indicate stronger ability in discriminating the pitch between two tones.
Change in Accuracy in Processing Rapid Presentation of Two Tones | Before & after 8-week intervention program
  Measures the change in the participants' ability in processing two rapid tones using the Rapid Auditory Processing task. The participant will be tested before intervention and after intervention. Two complex tones with fundamental frequency of 100Hz (Low tone) and 305Hz (High tone), each 75ms in duration, will be used throughout the entire test. For each trial, the participant will listen to two tones at ISI of 4ms, 8ms, or 30ms. The participants will be required to replicate the sequence of High or Low tones in each trial as quickly as possible. The accuracy of replicating the sequence will be used to assess the participants' ability.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Lui, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Centre of Learning Science, Kowloon Tong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymous individual participant data will be uploaded to an publicly accessible database should the results were published as a journal article.
Time Frame: Data will be provided when a journal article is published for indefinite time
Access Criteria: Access to the data will be made public. The link to the database will be provided in the journal article.

REFERENCES:
- [Background] Ashwin C, Baron-Cohen S, Wheelwright S, O'Riordan M, Bullmore ET. Differential activation of the amygdala and the 'social brain' during fearful face-processing in Asperger Syndrome. Neuropsychologia. 2007 Jan 7;45(1):2-14. doi: 10.1016/j.neuropsychologia.2006.04.014. Epub 2006 Jun 30. PMID 16806312
- [Background] Baron-Cohen S, Leslie AM, Frith U. Does the autistic child have a "theory of mind"? Cognition. 1985 Oct;21(1):37-46. doi: 10.1016/0010-0277(85)90022-8. No abstract available. PMID 2934210
- [Background] Bonnel A, Mottron L, Peretz I, Trudel M, Gallun E, Bonnel AM. Enhanced pitch sensitivity in individuals with autism: a signal detection analysis. J Cogn Neurosci. 2003 Feb 15;15(2):226-35. doi: 10.1162/089892903321208169. PMID 12676060
- [Background] Boucher J, Lewis V, Collis GM. Voice processing abilities in children with autism, children with specific language impairments, and young typically developing children. J Child Psychol Psychiatry. 2000 Oct;41(7):847-57. PMID 11079427
- [Background] Oram Cardy JE, Flagg EJ, Roberts W, Brian J, Roberts TP. Magnetoencephalography identifies rapid temporal processing deficit in autism and language impairment. Neuroreport. 2005 Mar 15;16(4):329-32. doi: 10.1097/00001756-200503150-00005. PMID 15729132
- [Background] Castelli F, Happe F, Frith U, Frith C. Movement and mind: a functional imaging study of perception and interpretation of complex intentional movement patterns. Neuroimage. 2000 Sep;12(3):314-25. doi: 10.1006/nimg.2000.0612. PMID 10944414
- [Background] Demopoulos C, Hopkins J, Kopald BE, Paulson K, Doyle L, Andrews WE, Lewine JD. Deficits in auditory processing contribute to impairments in vocal affect recognition in autism spectrum disorders: A MEG study. Neuropsychology. 2015 Nov;29(6):895-908. doi: 10.1037/neu0000209. Epub 2015 May 25. PMID 26011112
- [Background] Demopoulos C, Lewine JD. Audiometric Profiles in Autism Spectrum Disorders: Does Subclinical Hearing Loss Impact Communication? Autism Res. 2016 Jan;9(1):107-20. doi: 10.1002/aur.1495. Epub 2015 May 11. PMID 25962745
- [Background] Devine RT, Hughes C. Silent films and strange stories: theory of mind, gender, and social experiences in middle childhood. Child Dev. 2013 May-Jun;84(3):989-1003. doi: 10.1111/cdev.12017. Epub 2012 Nov 30. PMID 23199139
- [Background] Gaab N, Gabrieli JD, Deutsch GK, Tallal P, Temple E. Neural correlates of rapid auditory processing are disrupted in children with developmental dyslexia and ameliorated with training: an fMRI study. Restor Neurol Neurosci. 2007;25(3-4):295-310. PMID 17943007
- [Background] Gebauer L, Skewes J, Horlyck L, Vuust P. Atypical perception of affective prosody in Autism Spectrum Disorder. Neuroimage Clin. 2014 Oct 5;6:370-8. doi: 10.1016/j.nicl.2014.08.025. eCollection 2014. PMID 25379450
- [Background] Globerson E, Amir N, Kishon-Rabin L, Golan O. Prosody recognition in adults with high-functioning autism spectrum disorders: from psychoacoustics to cognition. Autism Res. 2015 Apr;8(2):153-63. doi: 10.1002/aur.1432. Epub 2014 Nov 26. PMID 25428545
- [Background] Golan O, Baron-Cohen S, Hill JJ, Golan Y. The "reading the mind in films" task: complex emotion recognition in adults with and without autism spectrum conditions. Soc Neurosci. 2006;1(2):111-23. doi: 10.1080/17470910600980986. PMID 18633780
- [Background] Grossman RB, Tager-Flusberg H. "Who said that?" Matching of low- and high-intensity emotional prosody to facial expressions by adolescents with ASD. J Autism Dev Disord. 2012 Dec;42(12):2546-57. doi: 10.1007/s10803-012-1511-2. PMID 22450703
- [Background] Hudepohl MB, Robins DL, King TZ, Henrich CC. The role of emotion perception in adaptive functioning of people with autism spectrum disorders. Autism. 2015 Jan;19(1):107-12. doi: 10.1177/1362361313512725. Epub 2013 Dec 11. PMID 24335115
- [Background] Jones CR, Happe F, Baird G, Simonoff E, Marsden AJ, Tregay J, Phillips RJ, Goswami U, Thomson JM, Charman T. Auditory discrimination and auditory sensory behaviours in autism spectrum disorders. Neuropsychologia. 2009 Nov;47(13):2850-8. doi: 10.1016/j.neuropsychologia.2009.06.015. Epub 2009 Jun 21. PMID 19545576
- [Background] Kamio Y, Inada N, Koyama T. A nationwide survey on quality of life and associated factors of adults with high-functioning autism spectrum disorders. Autism. 2013 Jan;17(1):15-26. doi: 10.1177/1362361312436848. Epub 2012 Mar 7. PMID 22399449
- [Background] Jones CR, Pickles A, Falcaro M, Marsden AJ, Happe F, Scott SK, Sauter D, Tregay J, Phillips RJ, Baird G, Simonoff E, Charman T. A multimodal approach to emotion recognition ability in autism spectrum disorders. J Child Psychol Psychiatry. 2011 Mar;52(3):275-85. doi: 10.1111/j.1469-7610.2010.02328.x. Epub 2010 Oct 18. PMID 20955187
- [Background] Kargas N, Lopez B, Reddy V, Morris P. The relationship between auditory processing and restricted, repetitive behaviors in adults with autism spectrum disorders. J Autism Dev Disord. 2015 Mar;45(3):658-68. doi: 10.1007/s10803-014-2219-2. PMID 25178987
- [Background] LaCava PG, Rankin A, Mahlios E, Cook K, Simpson RL. A single case design evaluation of a software and tutor intervention addressing emotion recognition and social interaction in four boys with ASD. Autism. 2010 May;14(3):161-78. doi: 10.1177/1362361310362085. Epub 2010 May 20. PMID 20488823
- [Background] Lerner MD, McPartland JC, Morris JP. Multimodal emotion processing in autism spectrum disorders: an event-related potential study. Dev Cogn Neurosci. 2013 Jan;3:11-21. doi: 10.1016/j.dcn.2012.08.005. Epub 2012 Sep 1. PMID 23245216
- [Background] Levitt H. Transformed up-down methods in psychoacoustics. J Acoust Soc Am. 1971 Feb;49(2):Suppl 2:467+. No abstract available. PMID 5541744
- [Background] Lindner JL, Rosen LA. Decoding of emotion through facial expression, prosody and verbal content in children and adolescents with Asperger's syndrome. J Autism Dev Disord. 2006 Aug;36(6):769-77. doi: 10.1007/s10803-006-0105-2. PMID 16639533
- [Background] Lyons M, Schoen Simmons E, Paul R. Prosodic development in middle childhood and adolescence in high-functioning autism. Autism Res. 2014 Apr;7(2):181-96. doi: 10.1002/aur.1355. Epub 2014 Mar 14. PMID 24634421
- [Background] Marshall CM, Snowling MJ, Bailey PJ. Rapid auditory processing and phonological ability in normal readers and readers with dyslexia. J Speech Lang Hear Res. 2001 Aug;44(4):925-40. doi: 10.1044/1092-4388(2001/073). PMID 11521783
- [Background] Moors A, De Houwer J. Automaticity: a theoretical and conceptual analysis. Psychol Bull. 2006 Mar;132(2):297-326. doi: 10.1037/0033-2909.132.2.297. PMID 16536645
- [Background] Ramdoss S, Machalicek W, Rispoli M, Mulloy A, Lang R, O'Reilly M. Computer-based interventions to improve social and emotional skills in individuals with autism spectrum disorders: a systematic review. Dev Neurorehabil. 2012;15(2):119-35. doi: 10.3109/17518423.2011.651655. PMID 22494084
- [Background] Taylor LJ, Maybery MT, Grayndler L, Whitehouse AJ. Evidence for shared deficits in identifying emotions from faces and from voices in autism spectrum disorders and specific language impairment. Int J Lang Commun Disord. 2015 Jul;50(4):452-66. doi: 10.1111/1460-6984.12146. Epub 2015 Jan 14. PMID 25588870
- [Background] Rutherford MD, Baron-Cohen S, Wheelwright S. Reading the mind in the voice: a study with normal adults and adults with Asperger syndrome and high functioning autism. J Autism Dev Disord. 2002 Jun;32(3):189-94. doi: 10.1023/a:1015497629971. PMID 12108620
- [Background] Santos A, Joly-Pottuz B, Moreno S, Habib M, Besson M. Behavioural and event-related potentials evidence for pitch discrimination deficits in dyslexic children: improvement after intensive phonic intervention. Neuropsychologia. 2007 Mar 14;45(5):1080-90. doi: 10.1016/j.neuropsychologia.2006.09.010. Epub 2006 Nov 30. PMID 17140611
- [Background] Schirmer A, Kotz SA. Beyond the right hemisphere: brain mechanisms mediating vocal emotional processing. Trends Cogn Sci. 2006 Jan;10(1):24-30. doi: 10.1016/j.tics.2005.11.009. PMID 16321562
- [Background] Stewart ME, McAdam C, Ota M, Peppe S, Cleland J. Emotional recognition in autism spectrum conditions from voices and faces. Autism. 2013 Jan;17(1):6-14. doi: 10.1177/1362361311424572. Epub 2012 Oct 8. PMID 23045218
- [Background] Wiethoff S, Wildgruber D, Kreifelts B, Becker H, Herbert C, Grodd W, Ethofer T. Cerebral processing of emotional prosody--influence of acoustic parameters and arousal. Neuroimage. 2008 Jan 15;39(2):885-93. doi: 10.1016/j.neuroimage.2007.09.028. Epub 2007 Sep 22. PMID 17964813